CLINICAL TRIAL: NCT01459081
Title: Randomised, Double-blind, Placebo-controlled Trial of Inhaled Zanamivir in Treatment of Influenza A and B Virus Infections in China
Brief Title: Efficacy and Safety of Inhaled Zanamivir in Treatment of Influenza A and B Virus Infections in China
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIM-100
Record Dates: First submitted 2011-10-21; First posted 2011-10-25 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Influenza A Virus Infection; Influenza B Virus Infection
MeSH Terms: interventions — Zanamivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zanamivir (Experimental)
  Interventions: Drug: Zanamivir
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zanamivir — 10 mg inhaled by mouth, twice daily, for 5 days
  Arms: Zanamivir
Drug: Placebo — inhaled by mouth, twice daily, for 5 days
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the clinical efficacy and safety of inhaled zanamivir in treatment of influenza A and B virus infections in China.

ELIGIBILITY:
Inclusion Criteria:

* Who had fever (>38.0ºC)
* At least two of the following symptoms: chills, headache, myalgia, fatigue, nasal symptoms, sore throat, cough
* Started therapy within 48 hours of onset of influenza-like illness
* Written informed consent

Exclusion Criteria:

* Respiratory diseases, such as asthma or COPD
* Woman with a positive urine pregnancy test
* Woman without contraception during the study
* Allergic to zanamivir, Paracetamol or lactose
* WBC ≥ 10.5×109/L; neutrophil percentage ≥ 80%
* Hepatic function impairment: AST ≥ 2×ULN, ALT ≥ 2×ULN
* Renal function impairment: Cr > 221μmol/L
* Influenza vaccination in the 12 months prior the beginning of the study
* History of tumor, psychiatric disorders, epilepsy or drug abuse
* Patients receiving corticosteroids, immunosuppressants
* HIV positive

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2011-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Time to alleviation of clinically important symptoms | up to 21 days

SECONDARY OUTCOMES:
Symptom score AUC | 6 days
Mean symptom scores | 6 days
The use of relief medication | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Qingyu Xiu, MD, Principal Investigator — Shanghai Changzheng Hospital
Locations (12):
- China (12):
  - The Third Xiangya Hospital Of Central South University, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - The First People's Hospital of Hangzhou, Hangzhou
  - The Affiliated Hospital of Inner Mongolia Medical College, Hohhot
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing
  - Qingdao Municipal Hospital, Qingdao
  - Shanghai 6th People's Hospital, Shanghai
  - Shanghai Changzheng Hospital, Shanghai
  - ShengJing Hospital of China Medical University, Shenyang
  - Tangdu Hospital Affiliated to the Fourth Military Medical University, Xi'an
  - Northern Jiangsu People's Hospital, Yangzhou